CLINICAL TRIAL: NCT06980168
Title: Effectiveness of Kabat Technique Verses Neural Mobilization With Facial Exercises in Bells Palsy
Brief Title: Kabat Technique vs Neural Mobilization in Bells Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-GCUF-079296
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Bell Palsy
Keywords: Facial nerve; Rehabilitation; Exercise therapy; Bell palsy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kabat technique (Active Comparator): kabat rehabilitation technique with baseline treatment
  Interventions: Other: kabat technique
- facial neural mobilization (Experimental): facial nerve mobilization with facial exercises
  Interventions: Other: facial nerve mobilization

INTERVENTIONS:
Other: kabat technique — kabat technique include diagonal movements to activate weak muscles through resistance . 3-5 repetetion per muscle for 2-3 sets .session conducted 5 days per week for three weeks each lasting 30 minutes .
  Arms: kabat technique
Other: facial nerve mobilization — neural mobilization involves manual traction and circular movement around ear to enhance nerve mobility and function .5-10 repetetions .Session conduted 5 days per week for 3 weeks lasting 30 minutes facial exercises include raising eyebrows-eye closure-lip raising-smiling-snarling flaring of nose-forehead wrinkling-lipspuckering-pouting. 5-10 repetetions 3 times a day .7 days for 3 weeks
  Arms: facial neural mobilization

SUMMARY:
The goal of this study is to compare the effect of kabat technique and neural mobilization with facial exercises in improving functional outcomes of patient with bells palsy

DETAILED DESCRIPTION:
Bells palsy is seventh cranial nerve disorder which causes muscle weaknesss on one side of the face .Various approaches are applied to restore facial function but this study aims to distinguish kabat technique and neural mobilization .This study will assess and compare the functional recovery of facial muscles and improvemrnt in facial symmetry .This will help determine which intervention is more effective .

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with bells palsy in less than 2 weeks

Exclusion Criteria:

* head injuries recent surgeries psycological issues multiple sclerosis

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
House-Brackman scale | 3rd week
  Changes from baseline in the House-Brackman scale will be used to assess the facial nerve dysfuntion. The tool grades facial movement on a scale from grade 1 to 6 where grade 1 indicates normal function and grade 6 indicates complete paralysis

SECONDARY OUTCOMES:
Facial disability index | 3rd week
  changes from baseline Facial disability index scores were assessed to determine functional improvement in facial movement. The FDI consists of two subscales physical function (5 items ) and socal function (5 items). Each item is scored individually and transformed to a scale of 0-100 with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoor Hassan, MS, Principal Investigator — Elite College of Management Science
Locations (1):
- Al raee hospital gujranwala ,Sardar yasin malik hospital, Rahat abdul gaffar medical complex, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No